CLINICAL TRIAL: NCT04430959
Title: A Pilot, Proof of Concept, Placebo-controlled Trial of Candesartan as an Adjunctive Treatment for Bipolar Depression
Brief Title: Candesartan as an Adjunctive Treatment for Bipolar Depression
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The reason the study was withdrawn was due to lack of funds. In addition, the PI is moving to a different institution and it would not be feasible to proceed with the study under these circumstances.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Marsal Sanches, Associate Director, UT Health Center of Excellence on Mood Disorders, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-19-1046
Record Dates: First submitted 2020-05-11; First posted 2020-06-16 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Bipolar Disorder Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Candesartan first then Placebo (Experimental): 4 weeks of candesartan with crossover to the other.
  Interventions: Drug: Candesartan; Drug: Placebo
- Placebo first then Candesartan (Placebo Comparator): 4 weeks of placebo with crossover to the other.
  Interventions: Drug: Candesartan; Drug: Placebo

INTERVENTIONS:
Drug: Candesartan — Candesartan 4 mg, tablets, orally, once daily for 4 weeks
  Other Names: Atacand
Drug: Placebo — Candesartan placebo-matching tablets, orally, once daily for 4 weeks

SUMMARY:
This study will assess the safety and tolerability of Candesartan when used in patients with Bipolar Disorder, in addition to their medication treatment.

DETAILED DESCRIPTION:
Pharmacological options for the treatment of Bipolar disorder (BD) are limited and a large proportion of patients does not show adequate response to treatment, especially in the case of bipolar depression. It has been hypothesized that dysfunctions in the renin-angiotensin system (RAS) may be involved in the pathophysiology of BD. We propose a double-blind, randomized, placebo-controlled, cross-over, proof-of-concept trial to investigate the effects of candesartan, an angiotensin-II receptor antagonist capable to cross the blood-brain barrier, as an adjunctive agent in the treatment of bipolar depression. Bipolar patients on a depressive episode will be randomly assigned to undergo two consecutive 4-week treatment periods with either candesartan (4 mg daily) or placebo in a crossover study. At the beginning of each treatment period, participants will complete a resting-state functional MRI scan, to be performed 1.5 hours after the first dose of the study medication. Subjects will be followed weekly and the Montgomery-Asberg Depression Rating Scale (MADRS) will be adopted as the primary outcome measure. Response will be defined as a decrease equal or higher than 50% in the MADRS score from the time of study entry to the 4th week of each treatment period. Possible associations between changes in brain connectivity (measured through resting state functional MRI) and subsequent response to treatment will also be analyzed.

ELIGIBILITY:
A diagnosis of BD type I or II, and currently in a depressive episode, based on DSM-5 criteria.

Inclusion criteria:

1. Age 18 to 65 years.
2. A diagnosis of BD type I or II according to DSM-5 criteria, established through the administration of the MINI.
3. Currently in a depressive episode, based on DSM-5 criteria.
4. MADRS >20 at entry in the study.
5. No history of hypertension, diabetes, stroke, liver, kidney, heart disease, bleeding disorders, cancer, hypothyroidism, auto-immune diseases, and any brain disorder (seizure disorder, stroke, dementia, or neurodegenerative diseases), as well as other conditions that could impact patient's safety associated with participation in the study.
6. On therapeutic doses of a mood stabilizing drug (anticonvulsants or atypical antipsychotics, but not lithium) or combinations of medications (including antidepressants, as long as receiving at least one mood stabilizing agent) for at least two weeks.
7. Allowed psychiatric comorbid conditions, such as anxiety disorders, PTSD and past history of substance use (as long as do NOT meet abuse or dependence criteria according to the SCID-I in the past 2 months).

Exclusion criteria:

1. Current use of angiotensin receptor antagonists, angiotensin converting enzyme inhibitors. (ACE inhibitors), or a history of allergies or poor tolerability to those medications
2. Current use of lithium or any other medications that could implicate in potentially dangerous. interactions with candesartan, based on available literature and the investigator's judgement.
3. Pregnancy or current breastfeeding.
4. Acute systemic infections or other acute medical conditions at the time of study entry.
5. Acute suicidal or homicidal ideation or other imminent concerns about safety, based on the investigator's judgement and/or on a score equal or higher than 4 in the item 10 of the MADRS.
6. Family history of hereditary neurologic disorder.
7. Unable to give informed consent for any reason.
8. Floating metallic objects in the body.
9. Positive urine drug screening at the time of study entry.
10. Current or previous diagnosis of intellectual disability, learning disability, or other severe neurodevelopmental disorders.
11. History of traumatic brain injury or head trauma with loss of consciousness for more than 30 minutes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) scores at the end of each treatment period. | Four weeks
  MADRS scores range from 0-60; higher scores indicate a higher level of severity of depressive symptoms. Response will be defined as a decrease equal or higher than 50% in the total MADRS score between the baseline and the 4th week of each treatment period.

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) scores at the end of each treatment period. | Four weeks
  HAM-A scores range from 0-56, with higher scores indicating more severe anxiety
Clinical Global Impression - Severity scale (CGI-S) scores at the end of each treatment period. | Four weeks
  The CGI-S is a 7-point scale used to rate the severity of the patient's illness at the time of assessment, compared to the clinician's past experience regarding patients with similar diagnosis
Functional Assessment Screening Tool scores at the end of each treatment period. | Four weeks
  The Functional Assessment Screening Tool (FAST) identifies factors that may influence problem behaviors. It is a self-report checklist that contains 16 items, with each questions being marked as either "yes", "no", or "not applicable". The checklist is designed to identify whether maladaptive behavior is maintained in four domains: attention/preferred items, escape from tasks/activities, sensory stimulation, pain attenuation.
Young Mania Rating Scale (YMRS) at the end of each treatment period | Four weeks
  The YMRS is one of the most frequently utilized rating scales to assess manic symptoms. The scale has 11 items, based on the patient's subjective report and observations made during the clinical interview. Higher scores indicate a greater severity of manic symptoms. Given the cyclic nature of BD, the YMRS will be utilized to monitor patients as for the possibility of a manic switch over each four-week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Marsal Sanches, MD PhD, Principal Investigator — University of Texas, Science Center at Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States